CLINICAL TRIAL: NCT02570529
Title: Prevention of Upper Gastrointestinal Hemorrhage Using Albis® in the Patients of Locally Advanced Pancreatic Cancer Who Underwent Concurrent Chemoradiotherapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator decided to stop the study because it was difficult to proceed with the study.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2015-0679
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic cancer; Chemoradiotherapy; Gastrointestinal toxicity; Albis
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albis® (Experimental): The intervention group
  Interventions: Drug: Albis®
- Placebo (Placebo Comparator): The placebo comparator group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albis® — The patients take Albis® 2T orally twice a day during the period between start day of concurrent chemoradiotherapy and 1 month after the treatment. During the period receiving radiation, the patient are prescribed the medication by the 2 weeks, and after radiation, they receive the 1 month's medication.
  Arms: Albis®
Drug: Placebo — The patients take placebo 2T orally twice a day during the period between start day of concurrent chemoradiotherapy and 1 month after the treatment. During the period receiving radiation, the patient are prescribed the medication by the 2 weeks, and after radiation, they receive the 1 month's medication.
  Arms: Placebo

SUMMARY:
Pancreatic ductal adenocarcinoma is the fourth cause of death in the Western world. About 40% of pancreatic cancer patients were diagnosed as locally advanced unresectable status without distant metastasis. Concurrent chemoradiotherapy (CCRT) was a reasonable treatment modality for locally advanced pancreatic cancer. However, several adverse events of chemoradiation could lead unfavorable treatment results, which included unique gastrointestinal (GI) toxicities, such as ulcer and hemorrhage in the stomach and duodenum that are included in the radiation field. According to the study in the investigators hospital, 45% of locally advanced pancreatic cancer patients treated with CCRT suffered from GI ulcers, and among them, 65% of the patients experienced the significant hemorrhage events. Although these GI toxicities, the studies for radioprotective agents were limited. Albis® is a newly developed drug comprised of ranitidine, bismuth and sucralfate. The investigators will investigate the radioprotective effect of Albis® for locally advanced pancreatic cancer patients treated with CCRT.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old and younger than 80 years old
* Pathologically confirmed pancreatic ductal adenocarcinoma (metastatic or locally advanced stage)
* ECOG Performance status ≤2
* Scheduled fot concurrent chemoradiation
* Adequate liver function (total bilirubin < 1.5 X the upper limits of normal (ULN), AST and ALT <3 X UNL, and alkaline phosphatases < 3 X ULN or < 5 x ULN in case of liver involvement)
* Adequate BM function (WBC ≥ 3,500/µl, absolute neutrophil cell count ≥ 1,500 /µl, platelet count ≥ 100,000/µl)
* Not remarkable coagulation profile (PT < 1.5 international normalized ratio(INR), aPTT <35 sec)
* Subjects who given written informed consent after being given a full description of the study

Exclusion Criteria:

* Coexisting of other malignancies within 5 years, except squamous cell carcinoma and basal cell carcinoma of the skin
* Evidence of distant metastasis, such as liver, peritoneum and brain
* history of receiving the chemoradiation for pancreatic cancer in the other hospital
* History of receiving the operation which affect the anatomy of upper gastrointestinal tract
* Any trouble for examination of upper endoscopy
* Evidence of GI ulcers (A1~H2) on endoscopy before start of chemoradiotherapy.
* Use of aspirin, anti-platelet agent, anticoagulation agent, NSAIDs, or glucocorticoid within 1 week or enable to stop the administration (including start during chemoradiation)
* Use of PPI, Histamine-2 receptor antagonist, antacid, prostaglandin, sucralfate within 2 weeks or enable to stop the administration
* Patients who are unwilling or unable to provide informed consent, such as those with psychiatric problem, drug abuse or alcoholism

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal ulcer incidence | within 4 weeks from end of chemoradiation
  After 1 month after the chemoradiation, all the patients receive the esophagogastroduodenoscopy to detect the development of gastrointestinal ulcers. The proportion of patients with radiation-induced GI ulcers in each group will be investigated

SECONDARY OUTCOMES:
Adverse event of gastrointestinal hemorrhage | within 4 weeks